CLINICAL TRIAL: NCT06025669
Title: Effects of Nap Restriction on Preschoolers' Empathy, Prosocial Behaviors and Executive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guanghai Wang, Developing Brain Lab, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCMCIRB-K2022122-2
Record Dates: First submitted 2023-08-07; First posted 2023-09-06 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Sleep Restriction
Keywords: nap restriction; preschooler; socio-emotional development; executive function; event-related potential

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nap rested and nap restriction (Experimental): There are two conditions in the single-arm, that is, the nap rested condition and the nap restriction condition. The sequence of two conditions is randomized.
  Interventions: Behavioral: Nap restriction

INTERVENTIONS:
Behavioral: Nap restriction — There are 2 interventions in the single-arm, that is, the nap rested condition and the nap restriction condition. The sequence of nap intervention followed randomization.

SUMMARY:
Cross-sectional evidences suggest a relationship between early childhood sleep and cognitive as well as socio-emotional functions. However, the casual relation has not been fully revealed. The current study aims to perform a randomized lab-based crossover nap restriction study on preschoolers, to determine the effects of sleep restriction on preschoolers empathy, prosocial behaviors as well as executive functions.

DETAILED DESCRIPTION:
The study will enroll preschoolers with regular nap habits. Under a randomized repeated-measures crossover design, they follow a strict sleep schedule (≥ 12.5 hours' time in bed every 24 hours) for 5 days, before each of two pseudorandomly assigned afternoon assessments following nap-rested or nap-restricted conditions. Actigraphy is applied to monitor sleep, and occipital alpha power is detected from resting-state EEG to objectively measure sleepiness. Empathy (Empathic for Pain Event-related Potential Paradigm) and prosocial behaviors (Concern for Others Behavioral Paradigm) were measured at each assessment. The effects of nap restriction were analyzed with paired t-test/Wilcoxon matched-pairs sign rank test and repeated-measures ANOVA.

ELIGIBILITY:
Inclusion Criteria:

1. healthy, typically developing, Intelligence quotient (IQ) ≥ 85;
2. never diagnosed with emotional-behavioral problems;
3. sleeping on a regular daily schedule;
4. reported napping three or more times every week, ≤ one nap in one day;
5. able to fall asleep by themselves.

Exclusion Criteria:

1. not able to fall asleep alone;
2. travel beyond two time zones within 3 months of the study;
3. use of medications influencing sleep or alertness;
4. reported or diagnosed sleep problems (such as obstructive sleep apnea (OSA), narcolepsy, parasomnia, insomnia, etc.) ;
5. history of neurodevelopmental diseases, including developmental delay, epilepsy, chronic medical conditions, lead poisoning and head injuries involving loss of consciousness;
6. conceptual age <35 weeks or > 45 weeks;
7. birth weight < 2,500 grams;
8. Children's Behaviors Checklist (CBCL) total score > 70;
9. a first-degree family history of diagnosed narcolepsy, psychosis or bipolar disorder.

Ages: 42 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Voltage of N2 and Late Positive Potential (LPP) components | 20 minutes after waking up from scheduled nap, or 20 minutes post nap restriction
  Child brain electroencephalogram (EEG) signals were collected via a non-invasive electrical brain cap and a wireless signal amplifier during the Empathic for Pain Event-related Potential Paradigm. The paradigm presents 32 pairs of empathic pain-related pictures at each sleep intervention condition (e.g., a hand hit by a hammer). The children are asked to think about "How painful do you think the person in the picture feels?" while looking at each picture. After data processing, the voltages of N2 (i.e. the negative potential at approximately 200 ms poststimulus) and LPP (a protracted slow-wave component elicited by emotional stimuli) are output and compared across sleep conditions.
Empathic pain rating | 20 minutes after waking up from scheduled nap, or 20 minutes post nap restriction
  The Empathic for Pain Event-related Potential Paradigm presents 32 pairs of empathic pain-related pictures at each sleep intervention condition (e.g., a hand hit by a hammer). The children are asked to rate on "How pain do you think the person in the picture feels?" with the Wong-Baker FACES Pain Rating System. The Wong-Baker FACES Pain Rating System includes 6 faces demonstrating painful expressions, scoring 0, 2, 4, 6, 8, and 10 points respectively, with higher scores representing higher levels of vicarious painful feelings. The mean scores of ratings are used to compare the empathy behavioral level across sleep conditions.

SECONDARY OUTCOMES:
Executive function - behavior | 20 minutes after waking up from scheduled nap, or 20 minutes post nap restriction
  The Heart and Flower Paradigm is used to measure child executive function. The children are asked to press left button while seeing a heart in the middle of the screen, and to press the right button while seeing a flower in the middle of the screen. The correct rate and response time is used to compare the executive performance across sleep conditions.
Executive function - EEG signal | 20 minutes after waking up from scheduled nap, or 20 minutes post nap restriction
  The Heart and Flower Paradigm is used to measure child executive function. The children are asked to press left button while seeing a heart in the middle of the screen, and to press the right button while seeing a flower in the middle of the screen. And the EEG signal are collected simultaneously. The β/Θ ratio of EEG signal is used to compare executive brain functions across sleep conditions.
Emotional arousal | 20 minutes after waking up from scheduled nap, or 20 minutes post nap restriction
  During the Concern for Others Paradigm, the child's epidermal electricity level is measured at baseline and during the pain demonstration, and the differences between baseline and during the pain demonstration are used to compare the child's emotional arousal across sleep conditions.
Emotion regulation | 20 minutes after waking up from scheduled nap, or 20 minutes post nap restriction
  During the Concern for Others Paradigm, the child's respiratory sinus arrhythmia level is measured at baseline and during the pain demonstration, and the differences between baseline and during the pain demonstration are used to compare the child's emotion regulation across sleep conditions.
Prosocial behavior level | 20 minutes after waking up from scheduled nap, or 20 minutes post nap restriction
  After the Empathic for Pain Event-related Potential Paradigm and Heart and Flower Paradigm are finished. Prosocial behaviors are measured under the Concern for Others Paradigm. Children are introduced to a playroom, where the experimenter plays with the child and "accidentally" hurts herself. The experimenter then demonstrates pain for one minute under standard procedure. Children's behaviors and expressions are recorded, and coded in four aspects: prosocial behaviors (1 to 6 points, higher scores represent higher levels of prosocial behaviors); empathic concern (1 to 4 points, higher scores represent higher levels of empathic concern); hypothesis testing (1 to 4 points, higher scores represent higher levels of hypothesis testing); and avoidance (0 to 1 points, higher scores represent higher levels of avoidance).

CONTACTS AND LOCATIONS:
Overall Officials: Fan Jiang, PhD, Study Director — Shanghai Children's Medical Center; Guanghai Wang, PhD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Miller AL, Seifer R, Crossin R, Lebourgeois MK. Toddler's self-regulation strategies in a challenge context are nap-dependent. J Sleep Res. 2015 Jun;24(3):279-87. doi: 10.1111/jsr.12260. Epub 2014 Nov 13. PMID 25394169
- [Background] Rong T, Sun X, Zhang Z, Li W, Deng Y, Wang Z, Meng M, Zhu Q, Jiang Y, Zhao J, Zhang Y, Wang G, Jiang F. The association between sleep and empathy in young preschoolers: A population study. J Sleep Res. 2022 Aug;31(4):e13530. doi: 10.1111/jsr.13530. Epub 2021 Dec 13. PMID 34904310
- [Background] Decety J, Meidenbauer KL, Cowell JM. The development of cognitive empathy and concern in preschool children: A behavioral neuroscience investigation. Dev Sci. 2018 May;21(3):e12570. doi: 10.1111/desc.12570. Epub 2017 May 18. PMID 28523733
- [Background] Roth-Hanania R, Davidov M, Zahn-Waxler C. Empathy development from 8 to 16 months: early signs of concern for others. Infant Behav Dev. 2011 Jun;34(3):447-58. doi: 10.1016/j.infbeh.2011.04.007. Epub 2011 May 20. PMID 21600660
- [Background] Adam N, Blaye A, Gulbinaite R, Delorme A, Farrer C. The role of midfrontal theta oscillations across the development of cognitive control in preschoolers and school-age children. Dev Sci. 2020 Sep;23(5):e12936. doi: 10.1111/desc.12936. Epub 2020 Feb 12. PMID 31894624
- [Background] Berger RH, Miller AL, Seifer R, Cares SR, LeBourgeois MK. Acute sleep restriction effects on emotion responses in 30- to 36-month-old children. J Sleep Res. 2012 Jun;21(3):235-46. doi: 10.1111/j.1365-2869.2011.00962.x. Epub 2011 Oct 11. PMID 21988087